CLINICAL TRIAL: NCT02125552
Title: A Randomized Control Trial of Ultrasound Guided IV Access in the Pediatric Emergency Department
Brief Title: Ultrasound Guided IV Access in a Pediatric Emergency Department
Acronym: USgIV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13-010758
Record Dates: First submitted 2014-04-24; First posted 2014-04-29 (Estimated); Last update posted 2018-05-15 (Actual); Status verified 2018-05

CONDITIONS: Difficult Intravenous Access in Pediatrics
Keywords: vascular access device; ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound guided intravenous access (Experimental): This group will have their IV placed by ultrasound guidance.
  Interventions: Procedure: Ultrasound guidance
- Traditional intravenous access (Placebo Comparator): The patients randomized to traditional IV access will have their IVs placed by standard technique.
  Interventions: Procedure: Traditional intravenous access

INTERVENTIONS:
Procedure: Ultrasound guidance — The ultrasound machine will be used to guide intravenous line placement in patients randomized to the ultrasound guided intravenous line group
  Arms: Ultrasound guided intravenous access
Procedure: Traditional intravenous access — Placement by experienced nurse using standard IV techniques
  Other Names: Standard of Care arm
  Arms: Traditional intravenous access

SUMMARY:
The primary objective is to determine whether the use of ultrasound guidance compared to standard IV access improves the proportion of successful IV placement on a first attempt for children in a pediatric emergency department who have predicted difficult access by a validated score. Secondary objectives include determining whether ultrasound-guided IV access lowers the overall number of IV attempts and/or reduces time to IV access. The investigators will also examine the duration of IV access and any complications related to IV access in both the traditional and ultrasound guided IV access group.

DETAILED DESCRIPTION:
The proposed study is a randomized trial of ultrasound guided IV access compared to traditional IV access in patients determined to have difficult IV access based on the Difficult Intravenous Access (DIVA) scale. Patients enrolled in the study will be randomized to traditional IV access or ultrasound guided IV access. If randomized to ultrasound guided IV access, the IV will be placed under direct visualization. Following IV placement or when attempts at IV access have ceased, the patient and family will be asked to complete a series of questions related to their satisfaction regarding IV placement. The follow-up phase examining duration of the IV and any related complications will continue until the IV placed as part of the study has been removed.

ELIGIBILITY:
Inclusion Criteria:

* Emergency department patients ages 0-18 years
* Requiring IV access as determined by emergency department attending physician
* Predicted difficult IV access as defined by a revised DIVA score >3

Exclusion Criteria:

* Unstable patients triaged as a Level 1 triage acuity
* Patients who refuse IV access
* Non-English speaking parent/guardian
* No study team member available to enroll patient
* Parent/guardian does not consent
* Allergy to ultrasound gel

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 163 (Actual)
Dates: Start 2014-05; Primary Completion 2016-12-02 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Success of Initial IV Placement Attempt | Participants will be followed through the duration of emergency department stay, an expected average of 4 hours
  Patients will be randomized to traditional IV placement or ultrasound guided IV placement immediately after enrollment. The IV will be placed directly following enrollment.

SECONDARY OUTCOMES:
Measure the overall number of IV attempts.. | Participants will be followed through the duration of emergency department stay, an expected average of 4 hours
  We will record the number of IV attempts made until a patient has a successfully placed IV or further attempts are aborted.
Time to IV access. | Participants will be followed through the duration of emergency department stay, an expected average of 4 hours
  The time from enrollment until successful IV access is obtained will be measured.
Patient & family satisfaction with IV placement method. | Participants will be followed through the duration of emergency department stay, an expected average of 4 hours
  A survey will be given to parents and patients over age 12 years to ask them about their experience with the IV placement.
Compare the survival (in length of time) of IV access | Participants will be followed through the duration of hospital stay, expected average of 5 days
  We will track the IVs placed as part of the study through the electronic medical record to determine when and why they were removed and if there were any associated complications.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph J Zorc, MD, MSCE, Principal Investigator — Children's Hospital of Philadelphia
Locations (1):
- The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Fein JA, Callahan JM, Boardman CR, Gorelick MH. Predicting the need for topical anesthetic in the pediatric emergency department. Pediatrics. 1999 Aug;104(2):e19. doi: 10.1542/peds.104.2.e19. PMID 10429137
- [Background] Frey AM. Success rates for peripheral i.v. insertion in a children's hospital. Financial implications. J Intraven Nurs. 1998 May-Jun;21(3):160-5. PMID 9652275
- [Background] Yen K, Riegert A, Gorelick MH. Derivation of the DIVA score: a clinical prediction rule for the identification of children with difficult intravenous access. Pediatr Emerg Care. 2008 Mar;24(3):143-7. doi: 10.1097/PEC.0b013e3181666f32. PMID 18347490
- [Background] Riker MW, Kennedy C, Winfrey BS, Yen K, Dowd MD. Validation and refinement of the difficult intravenous access score: a clinical prediction rule for identifying children with difficult intravenous access. Acad Emerg Med. 2011 Nov;18(11):1129-34. doi: 10.1111/j.1553-2712.2011.01205.x. PMID 22092893
- [Background] Doniger SJ, Ishimine P, Fox JC, Kanegaye JT. Randomized controlled trial of ultrasound-guided peripheral intravenous catheter placement versus traditional techniques in difficult-access pediatric patients. Pediatr Emerg Care. 2009 Mar;25(3):154-9. doi: 10.1097/PEC.0b013e31819a8946. PMID 19262420
- [Background] Keyes LE, Frazee BW, Snoey ER, Simon BC, Christy D. Ultrasound-guided brachial and basilic vein cannulation in emergency department patients with difficult intravenous access. Ann Emerg Med. 1999 Dec;34(6):711-4. doi: 10.1016/s0196-0644(99)70095-8. PMID 10577399
- [Background] Au AK, Rotte MJ, Grzybowski RJ, Ku BS, Fields JM. Decrease in central venous catheter placement due to use of ultrasound guidance for peripheral intravenous catheters. Am J Emerg Med. 2012 Nov;30(9):1950-4. doi: 10.1016/j.ajem.2012.04.016. Epub 2012 Jul 15. PMID 22795988
- [Background] Gregg SC, Murthi SB, Sisley AC, Stein DM, Scalea TM. Ultrasound-guided peripheral intravenous access in the intensive care unit. J Crit Care. 2010 Sep;25(3):514-9. doi: 10.1016/j.jcrc.2009.09.003. Epub 2009 Oct 15. PMID 19836193
- [Background] Dargin JM, Rebholz CM, Lowenstein RA, Mitchell PM, Feldman JA. Ultrasonography-guided peripheral intravenous catheter survival in ED patients with difficult access. Am J Emerg Med. 2010 Jan;28(1):1-7. doi: 10.1016/j.ajem.2008.09.001. PMID 20006193
- [Background] Benkhadra M, Collignon M, Fournel I, Oeuvrard C, Rollin P, Perrin M, Volot F, Girard C. Ultrasound guidance allows faster peripheral IV cannulation in children under 3 years of age with difficult venous access: a prospective randomized study. Paediatr Anaesth. 2012 May;22(5):449-54. doi: 10.1111/j.1460-9592.2012.03830.x. Epub 2012 Mar 12. PMID 22409596
- [Background] Heinrichs J, Fritze Z, Vandermeer B, Klassen T, Curtis S. Ultrasonographically guided peripheral intravenous cannulation of children and adults: a systematic review and meta-analysis. Ann Emerg Med. 2013 Apr;61(4):444-454.e1. doi: 10.1016/j.annemergmed.2012.11.014. Epub 2013 Feb 15. PMID 23415740
- [Background] Bair AE, Rose JS, Vance CW, Andrada-Brown E, Kuppermann N. Ultrasound-assisted peripheral venous access in young children: a randomized controlled trial and pilot feasibility study. West J Emerg Med. 2008 Nov;9(4):219-24. PMID 19561750
- [Background] Aponte H, Acosta S, Rigamonti D, Sylvia B, Austin P, Samolitis T. The use of ultrasound for placement of intravenous catheters. AANA J. 2007 Jun;75(3):212-6. PMID 17591303
- [Background] Bauman M, Braude D, Crandall C. Ultrasound-guidance vs. standard technique in difficult vascular access patients by ED technicians. Am J Emerg Med. 2009 Feb;27(2):135-40. doi: 10.1016/j.ajem.2008.02.005. PMID 19371518
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Lininger RA. Pediatric peripheral i.v. insertion success rates. Pediatr Nurs. 2003 Sep-Oct;29(5):351-4. PMID 14651305
- [Background] Panebianco NL, Fredette JM, Szyld D, Sagalyn EB, Pines JM, Dean AJ. What you see (sonographically) is what you get: vein and patient characteristics associated with successful ultrasound-guided peripheral intravenous placement in patients with difficult access. Acad Emerg Med. 2009 Dec;16(12):1298-1303. doi: 10.1111/j.1553-2712.2009.00520.x. Epub 2009 Nov 12. PMID 19912132
- [Background] Schnadower D, Lin S, Perera P, Smerling A, Dayan P. A pilot study of ultrasound analysis before pediatric peripheral vein cannulation attempt. Acad Emerg Med. 2007 May;14(5):483-5. doi: 10.1197/j.aem.2006.12.016. PMID 17392522
- [Derived] Vinograd AM, Chen AE, Woodford AL, Fesnak S, Gaines S, Elci OU, Zorc JJ. Ultrasonographic Guidance to Improve First-Attempt Success in Children With Predicted Difficult Intravenous Access in the Emergency Department: A Randomized Controlled Trial. Ann Emerg Med. 2019 Jul;74(1):19-27. doi: 10.1016/j.annemergmed.2019.02.019. Epub 2019 May 22. PMID 31126618